CLINICAL TRIAL: NCT01656200
Title: A Prospective, Open Label Study of Human T Cell Responses to Live Attenuated Japanese Encephalitis Vaccine SA14-14-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indian Institute of Science (Other Government)
Collaborators: National Institute of Mental Health and Neuro Sciences, India (Other); University of Liverpool (Other); PATH (Other); Wellcome Trust (Other)
Responsible Party: Principal Investigator, Prof S Vijaya, Dr. Lance Turtle, Professor, Indian Institute of Science
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: JEV SA14-14-2/T cell/01
Record Dates: First submitted 2012-07-27; First posted 2012-08-02 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Japanese Encephalitis; Japanese Encephalitis Vaccine
Keywords: Japanese encephalitis; Japanese encephalitis vaccine; T lymphocyte; Immune response
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine (Experimental): Single dose live attenuated Japanese encephalitis vaccine SA14-14-2
  Interventions: Biological: Live attenuated Japanese encephalitis vaccine SA14-14-2

INTERVENTIONS:
Biological: Live attenuated Japanese encephalitis vaccine SA14-14-2 — Live attenuated Japanese encephalitis vaccine SA14-14-2

SUMMARY:
Japanese encephalitis (JE) live attenuated vaccine SA14-14-2 has been in use for more more than 20 years in Asia. JE vaccine SA14-14-2 is licensed in India and has been widely used since 2006. JE vaccines give protection by generating a neutralizing antibody response, but both naturally exposed persons and patients with JE also have T cell responses. Whether JE vaccine SA14-14-2 elicits T cell responses is unknown. This study tests the hypothesis that T cell responses are generated in response to JE SA14-14-2 vaccination. The aim of this study is to characterize T cell responses to JE vaccine SA14-14-2 in healthy people, and to investigate differences in T cell responses between natural exposure, vaccination and disease.

ELIGIBILITY:
Inclusion criteria:

* A male or female adult between 18 and 50 years of age.
* Written informed consent.
* Free of obvious health problems as established by medical history and history- directed physical examination before entering the study.
* Expected continuous residence in India during study period, without travel outside India
* An efficacious method of contraception must be used during the study for women of childbearing potential.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding administration of SA14-14-2 vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within a period of six months before vaccination or at any time during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition.
* A family history of congenital or hereditary immunodeficiency.
* Any antiviral drug therapy within a period of six months before vaccination or at any time during the study period.
* History of significant allergic disease or reactions likely to be exacerbated by any component of the study vaccine, especially allergic disease or reactions to any previous dose of any vaccine.
* History of having received JE vaccine, yellow fever vaccine, tick-borne encephalitis vaccine or experimental flavivirus vaccine.
* History of documented JE infection.
* Detectable anti JE or West Nile neutralizing antibodies in screening tests.
* Acute disease at the time of enrollment. Entry into the study may be deferred until the illness is resolved.
* Acute or chronic, clinically significant, pulmonary, cardiovascular, hepatic, neurological or renal functional abnormality, as determined by history and physical or laboratory examination that is not controlled by drugs.
* Administration of immunoglobulins and/or any blood products within the three months preceding administration of vaccine, or planned administration during the study period.
* Seropositive for HIV, HCV or HbsAg.
* Lactation, pregnancy or intention to get pregnant.
* History of excessive alcohol consumption, drug abuse or significant psychiatric illness.
* Any other condition that in the opinion of the investigator would pose a health risk to the participant or interfere with the evaluation of the vaccine.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof S Vijaya, PhD, Principal Investigator — Indian Institute of Science; Dr V Ravi, MBBS MD, Principal Investigator — National Institute of Mental Health and Neuro Sciences, India
Locations (2):
- India (2):
  - Indian Institute of Science, Bangalore, Karnataka
  - National Institute of Mental Health and Neurosciences, Bangalore, Karnataka

REFERENCES:
- [Derived] Turtle L, Tatullo F, Bali T, Ravi V, Soni M, Chan S, Chib S, Venkataswamy MM, Fadnis P, Yaich M, Fernandez S, Klenerman P, Satchidanandam V, Solomon T. Cellular Immune Responses to Live Attenuated Japanese Encephalitis (JE) Vaccine SA14-14-2 in Adults in a JE/Dengue Co-Endemic Area. PLoS Negl Trop Dis. 2017 Jan 30;11(1):e0005263. doi: 10.1371/journal.pntd.0005263. eCollection 2017 Jan. PMID 28135273

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaccine
Started | 17
Completed | 16
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Healthy South Indian Adults resident in Bengaluru, Karnataka State
Arm/Group | Vaccine
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 25 [20 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Region of Enrollment [Number; unit: Count of participants]
  India | 17

OUTCOME MEASURES:

1. Primary Outcome: Change of T Lymphocyte Responses to Live Attenuated JE SA-14-14-2 Vaccine at Week 2.
Description: Interferon gamma (IFNγ) spot forming cells (SFC)/million peripheral blood mononuclear cells (PBMC) at week 2 (peak response)
Time Frame: Week 1, week 2, week 4, week 8, 6 months
Population: 15 participants had data available at the two week time point. 1 withdrew beforehand, 1 declined to donate thew two week blood sample.
Measure: Geometric Mean (Full Range); unit: IFNγ SFC/million PBMC
Arm/Group | Vaccine
Number analyzed (Participants) | 15
IFNγ SFC/million PBMC | 34 [0 to 537]

2. Secondary Outcome: Neutralizing Antibody Titres to Live Attenuated JE SA-14-14-2 Vaccine at Week 4 Post Vaccination.
Description: Neutralizing antibody titres (measured by 50% Plaque reduction neutralisation titre (PRNT50)) at 4 weeks post vaccination
Time Frame: 4 weeks
Population: 1 participant withdrew before the 4 week time point, for another the sample was not available for analysis.
Measure: Geometric Mean (Full Range); unit: Neutralising antibody titres
Arm/Group | Vaccine
Number analyzed (Participants) | 15
Neutralising antibody titres | 18.5 [0 to 1188]

3. Secondary Outcome: Number of Participants Reporting Adverse Events (Graded in Severity 1-4).
Time Frame: one month
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine
Number analyzed (Participants) | 17
Participants | 3

ADVERSE EVENTS:
Arm/Group | Vaccine
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 3/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=17)
Fever, headache, myalgia, sore throat (General disorders) | 1 (1)
Fever, dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness, Headache (Nervous system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Dizziness for 2-3 seconds a time (Nervous system disorders) | 1 (1)
Fever, myalgia (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No